CLINICAL TRIAL: NCT01999218
Title: A Phase III, Multicenter, Randomized, Double-Blind, Active-Comparator-Controlled Clinical Trial to Study the Safety and Efficacy of the Addition of Ertugliflozin (MK-8835/PF-04971729) Compared With the Addition of Glimepiride in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin
Brief Title: Ertugliflozin vs. Glimepiride in Type 2 Diabetes Mellitus (T2DM) Participants on Metformin (MK-8835-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-002; 2013-003582-34 (EudraCT Number); B1521013 (Other: Pfizer)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Metformin; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertugliflozin 5 mg (Experimental): Ertugliflozin 5 mg once daily (QD) from Day 1 to Week 104
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to Ertugliflozin; Drug: Placebo to Glimepiride; Drug: Metformin; Drug: Sitagliptin
- Ertugliflozin 15 mg (Experimental): Ertugliflozin 15 mg QD from Day 1 to Week 104
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Ertugliflozin 10 mg; Drug: Placebo to Glimepiride; Drug: Metformin; Drug: Sitagliptin
- Glimepiride up to 8 mg (Active Comparator): Glimepiride to a maximum of 8 mg QD from Day 1 to Week 104
  Interventions: Drug: Glimerpiride; Drug: Placebo to Ertugliflozin; Drug: Metformin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin, 5 mg, oral, once daily, from Day 1 to Week 104
  Other Names: MK-8835
  Arms: Ertugliflozin 15 mg; Ertugliflozin 5 mg
Drug: Ertugliflozin 10 mg — Ertugliflozin, 10 mg, oral, once daily from Day 1 to Week 104.
  Other Names: MK-8355
  Arms: Ertugliflozin 15 mg
Drug: Glimerpiride — Glimepiride, oral tablets, initiated at 1 mg daily and titrated up to the maximum approved dose (8 mg daily based on the local country label) or maximum tolerated dose
  Arms: Glimepiride up to 8 mg
Drug: Placebo to Ertugliflozin — Matching placebo to ertugliflozin, 5 mg and/or 10 mg, oral, once daily, from Day 1 to Week 104
  Arms: Ertugliflozin 5 mg; Glimepiride up to 8 mg
Drug: Placebo to Glimepiride — Matching placebo to glimepiride, 1 mg or 2 mg, oral, once daily, from Day 1 to Week 104.
  Arms: Ertugliflozin 15 mg; Ertugliflozin 5 mg
Drug: Metformin — Participants are to remain on their stable doses of metformin (oral, >=1500 mg/day) while receiving blinded investigational product during the double-blind treatment period. Participants on metformin <1500 at screening are up-titrated to >= 1500 daily.
Drug: Sitagliptin — Open label, oral, once daily, rescue medication as required.

SUMMARY:
This study will evaluate the efficacy and safety of the addition of ertugliflozin (MK-8835/PF-04971729) compared with the addition of glimepiride in participants with T2DM who have inadequate glycemic control on metformin. The primary hypothesis of this study is that after 52 weeks, the change from baseline in hemoglobin A1c (A1C) in participants treated with the addition of ertugliflozin 15 mg once daily is non-inferior compared with that in participants treated with the addition of glimepiride.

DETAILED DESCRIPTION:
The duration of the trial will be up to approximately 122 weeks. This will include a 1-week screening period, an up to 13-week wash-off/titration/dose stabilization period, a 2-week placebo run-in period, a 104-week double-blind, active comparator-controlled treatment period, and a post-treatment telephone contact 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM in accordance to American Diabetes Association guidelines
* On metformin monotherapy or metformin in combination with a single allowable anti-hyperglycemic agent (AHA), DPP-4 inhibitors, meglitinides and AGIs are listed as allowable AHAs along with sulfonylureas prior to study participation.
* Body Mass Index (BMI) ≥18.0 kg/m^2
* Male or female not of reproductive potential
* If a female of reproductive potential, agree to remain abstinent or to use (or have their partner use) 2 acceptable combinations of birth control while participating in the trial and for 14 days after the last use of study drug.

Exclusion Criteria:

* History or presence of type 1 diabetes mellitus or a history of ketoacidosis
* History of other specific types of diabetes (eg, genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* A known hypersensitivity or intolerance to any sodium-glucose co-transporter 2 (SGLT2) inhibitor
* Use of the following prohibited therapeutic agents within 12 weeks of study participation: insulin, injectable anti-hyperglycemic agents, pioglitazone or rosiglitazone, another SGLT2 inhibitor, bromocriptine (Cycloset®), colesevelam (Welchol®), and any other non-approved anti-hyperglycemic therapy
* Known hypersensitivity or intolerance to metformin or glimepiride
* On a weight-loss program or medication or medication associated with weight changes and is not weight-stable (>=5% change in body weight in the last 6 months)
* History of bariatric surgery less than 12 months prior to study participation
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study participation
* Active, obstructive uropathy or an indwelling urinary catheter
* A history of malignancy ≤5 years prior to study participation, except for adequately treated basal or squamous cell skin cancer or in situ cervical cancer
* Known history of Human Immunodeficiency Virus (HIV)
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells
* A medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C (assessed by medical history), primary biliary cirrhosis, or symptomatic gallbladder disease
* Any clinically significant malabsorption condition
* Being treated for hyperthyroidism, or on thyroid replacement therapy that has not been at a stable dose for at least 6 weeks prior to study participation
* Previous randomization in a study with ertugliflozin
* Participation in other studies involving investigational drug(s) within 30 days of study participation and/or during the pre-randomization period
* A surgical procedure within 6 weeks prior to study participation or planned major surgery during the trial
* A positive urine pregnancy test
* Pregnant or breast-feeding, or expecting to conceive during the trial, including 14 days following the last dose of study drug
* Undergoing hormonal therapy in preparation to donate eggs during the period of the trial, including 14 days following the last dose of study drug
* Consumption of more than 2 alcoholic drinks per day or engages in binge drinking
* Donation of blood or blood products within 6 weeks of study participation or plans to donate blood or blood products at any time during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1326 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hollander P, Hill J, Johnson J, Wei Jiang Z, Golm G, Huyck S, Terra SG, Mancuso JP, Engel SS, Lauring B, Liu J. Results of VERTIS SU extension study: safety and efficacy of ertugliflozin treatment over 104 weeks compared to glimepiride in patients with type 2 diabetes mellitus inadequately controlled on metformin. Curr Med Res Opin. 2019 Aug;35(8):1335-1343. doi: 10.1080/03007995.2019.1583450. Epub 2019 Mar 25. PMID 30760125
- [Derived] Gallo S, Calle RA, Terra SG, Pong A, Tarasenko L, Raji A. Effects of Ertugliflozin on Liver Enzymes in Patients with Type 2 Diabetes: A Post-Hoc Pooled Analysis of Phase 3 Trials. Diabetes Ther. 2020 Aug;11(8):1849-1860. doi: 10.1007/s13300-020-00867-1. Epub 2020 Jul 9. PMID 32648108
- [Derived] Patel S, Hickman A, Frederich R, Johnson S, Huyck S, Mancuso JP, Gantz I, Terra SG. Safety of Ertugliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Seven Phase 3 Randomized Controlled Trials. Diabetes Ther. 2020 Jun;11(6):1347-1367. doi: 10.1007/s13300-020-00803-3. Epub 2020 May 5. PMID 32372382
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Wu L, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Efficacy and safety of ertugliflozin across racial groups in patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Aug;36(8):1277-1284. doi: 10.1080/03007995.2020.1760228. Epub 2020 May 13. PMID 32324082
- [Derived] Liu J, Tarasenko L, Pong A, Huyck S, Patel S, Hickman A, Mancuso JP, Ellison MC, Gantz I, Terra SG. Efficacy and safety of ertugliflozin in Hispanic/Latino patients with type 2 diabetes mellitus. Curr Med Res Opin. 2020 Jul;36(7):1097-1106. doi: 10.1080/03007995.2020.1760227. Epub 2020 May 13. PMID 32324065
- [Derived] Cherney DZI, Heerspink HJL, Frederich R, Maldonado M, Liu J, Pong A, Xu ZJ, Patel S, Hickman A, Mancuso JP, Gantz I, Terra SG. Effects of ertugliflozin on renal function over 104 weeks of treatment: a post hoc analysis of two randomised controlled trials. Diabetologia. 2020 Jun;63(6):1128-1140. doi: 10.1007/s00125-020-05133-4. Epub 2020 Mar 31. PMID 32236732
- [Derived] Liu J, Patel S, Cater NB, Wu L, Huyck S, Terra SG, Hickman A, Darekar A, Pong A, Gantz I. Efficacy and safety of ertugliflozin in East/Southeast Asian patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2020 Apr;22(4):574-582. doi: 10.1111/dom.13931. Epub 2020 Jan 3. PMID 31797522
- [Derived] Hollander P, Liu J, Hill J, Johnson J, Jiang ZW, Golm G, Huyck S, Terra SG, Mancuso JP, Engel SS, Lauring B. Ertugliflozin Compared with Glimepiride in Patients with Type 2 Diabetes Mellitus Inadequately Controlled on Metformin: The VERTIS SU Randomized Study. Diabetes Ther. 2018 Feb;9(1):193-207. doi: 10.1007/s13300-017-0354-4. Epub 2017 Dec 27. PMID 29282633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 16 countries at 232 trial centers in Argentina, Canada, Czech Republic, Hungary, South Korea, Lithuania, Mexico, Philippines, Poland, Romania, Russia, Slovakia, South Africa, Taiwan, Ukraine, and the United States.
Pre-assignment Details: A total of 1326 participants were randomized. Ten randomized participants from one trial site were excluded from all final analyses (Week 104 and beyond), and one randomized participant did not receive treatment.
Groups:
- Glimepiride: Glimepiride to a maximum of 8 mg QD from Day 1 to Week 104
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Started | 448 | 441 | 437
Treated | 448 | 440 | 437
Site Issue (Treated (excluding 1 trial site)) | 445 | 435 | 435
Completed | 339 | 340 | 327
Not Completed | 109 | 101 | 110
Not completed — Hyperglycemia | 18 | 17 | 17
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 22 | 17 | 18
Not completed — Non-Compliance With Study Drug | 6 | 4 | 1
Not completed — Physician Decision | 1 | 4 | 6
Not completed — Protocol Violation | 4 | 5 | 4
Not completed — Screen failure | 0 | 1 | 0
Not completed — Study Terminated By Sponsor | 7 | 5 | 12
Not completed — Participant moves | 2 | 5 | 3
Not completed — Withdrawal by Subject | 28 | 29 | 34
Not completed — Creatinine/eGFR | 0 | 0 | 1
Not completed — Death | 7 | 1 | 2
Not completed — Excluded Medication | 1 | 1 | 2
Not completed — Adverse Event | 9 | 7 | 7
Not completed — Treated but excluded at 1 trial site | 3 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride | Total
Number analyzed (Participants) | 448 | 441 | 437 | 1326
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All randomized participants
  Years | 58.8 (9.7) | 58.0 (9.9) | 57.8 (9.2) | 58.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — All randomized participants
  Participants
    Female | 221 | 250 | 213 | 684
    Male | 227 | 191 | 224 | 642
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All randomized participants
  Participants
    American Indian or Alaska Native | 5 | 3 | 5 | 13
    Asian | 81 | 86 | 73 | 240
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 17 | 19 | 25 | 61
    White | 332 | 316 | 318 | 966
    More than one race | 13 | 17 | 16 | 46
    Unknown or Not Reported | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: All randomized participants and treated participants.
  Kilograms
    number analyzed (Participants) | 448 | 440 | 437 | 1325
    (all) | 87.9 (18.9) | 85.6 (19.1) | 86.8 (20.7) | 86.8 (19.6)
Hemoglobin A1C [Mean (Standard Deviation); unit: Percentage] — Population: All randomized participants with a baseline A1C measurement.
  Percentage
    number analyzed (Participants) | 448 | 440 | 437 | 1325
    (all) | 7.81 (0.60) | 7.80 (0.60) | 7.76 (0.60) | 7.79 (0.60)
Sitting Systolic Blood Pressure [Mean (Standard Deviation); unit: Millimeters of mercury] — Population: All randomized participants with baseline sitting systolic blood pressure data.
  Millimeters of mercury
    number analyzed (Participants) | 448 | 440 | 437 | 1325
    (all) | 130.2 (12.8) | 130.8 (12.4) | 129.9 (12.0) | 130.3 (12.4)
Prior Antihyperglycemic (AHA) Medication (Monotherapy or Dual Therapy) [Count of Participants; unit: Participants] — Population: All randomized participants with information on or baseline data of prior antihyperglycemic medication use
  Participants
    Prior Antihyperglycemic Medication | 448 | 439 | 437 | 1324
    No Prior Use & Not on Antihyperglycemic Medication | 0 | 1 | 0 | 1
    Data not available | 0 | 1 | 0 | 1
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: milliliters/minute/1.73 meters^2] — Population: All randomized and treated participants.
  milliliters/minute/1.73 meters^2
    number analyzed (Participants) | 448 | 440 | 437 | 1325
    (all) | 88.3 (18.7) | 86.7 (18.3) | 86.6 (18.5) | 87.2 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 52: Excluding Rescue Approach
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). A1C represents the percentage of glycated hemoglobin. This change from baseline reflects the Week 52 A1C minus the Week 0 A1C. A negative number indicates a reduction in A1C level. Participants who met glycemic rescue criteria received open-label sitagliptin glycemic rescue medication. The primary study objective was the MK-8835 15 mg vs. glimepiride comparison; the MK-8835 5mg vs glimerpiride comparison was a secondary study objective.
Time Frame: Baseline and Week 52
Population: All randomized, treated participants with at least one A1C measurement (baseline or a post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 448 | 440 | 437
Percent | -0.56 [-0.65 to -0.47] | -0.64 [-0.73 to -0.55] | -0.74 [-0.83 to -0.65]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Non-Inferiority — Non-inferiority is declared if the upper bound of the two-sided 95% confidence interval (CI) for the mean difference is less than 0.3%; Difference in the Least Squares Means = 0.10, 95% CI 2-sided [-0.02 to 0.22] — Constrained Longitudinal Data Analysis (cLDA) model with fixed effects for treatment, time, prior antihyperglycemic medication (monotherapy or dual therapy), baseline eGFR (continuous) and the interaction of time by treatment
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in the Least Squares means = 0.18, 95% CI 2-sided [0.06 to 0.30] — Based on cLDA model with fixed effects for treatment, time, prior antihyperglycemic medication (monotherapy or dual therapy), baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable

2. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE) Up to Week 106
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Week 106
Population: All randomized participants who took at least one dose of trial treatment, 10 randomized participants from one trial site were excluded from these analyzes, and one randomized participant did not receive treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 445 | 435 | 435
Percentage of Participants | 70.1 | 71.3 | 69.7
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Other — Based on Miettinen & Nurminen method; Difference in % vs. Glimepiride = 1.6, 95% CI 2-sided [-4.5 to 7.7]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Other — Based on Miettinen & Nurminen method; Difference in % vs. Glimepiride = 0.5, 95% CI 2-sided [-5.6 to 6.5]

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE Up to Week 104
Description: as for outcome 2
Time Frame: Up to Week 104
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 445 | 435 | 435
Percentage of Participants | 6.5 | 8.0 | 5.1
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Other; Difference in % vs. Glimepiride = 3.0, 95% CI 2-sided [-0.3 to 6.4]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Other; Difference in % vs. Glimepiride = 1.5, 95% CI 2-sided [-1.7 to 4.7]

4. Secondary Outcome: Percentage of Participants With an Adverse Event of Symptomatic Hypoglycemia Up to Week 52: Excluding Rescue Approach
Description: Symptomatic hypoglycemia was an event with clinical symptoms reported by the investigator as hypoglycemia (biochemical documentation not required). Participants who met glycemic rescue criteria received open-label sitagliptin glycemic rescue medication.
Time Frame: Up to Week 52
Population: All randomized participants who took at least one dose of trial treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 448 | 440 | 437
Percentage of Participants | 3.1 | 5.2 | 19.2
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Other; p < 0.001, Based on Miettinen & Nurminen method; Difference in % vs. Glimepiride = -14.0, 95% CI 2-sided [-18.4 to -9.8]; Based on Miettinen & Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Other; p < 0.001, Based on Miettinen & Nurminen method; Difference in % vs. Glimepiride = -16.1, 95% CI 2-sided [-20.3 to -12.2]; Based on Miettinen & Nurminen method

5. Secondary Outcome: Change From Baseline in Body Weight at Week 52 Excluding Rescue Approach
Description: This change from baseline reflects the Week 52 body weight minus the Week 0 body weight. Participants who met glycemic rescue criteria received open-label sitagliptin glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: All randomized, treated participants with at least one body weight measurement (baseline or a post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 448 | 440 | 437
Kilograms | -2.96 [-3.31 to -2.61] | -3.38 [-3.73 to -3.03] | 0.91 [0.56 to 1.25]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Other; p < 0.001, Constrained Longitudinal Data analysis; Difference in LSM vs. Glimepiride = -4.29, 95% CI 2-sided [-4.77 to -3.80] — LSM=Least Squares Means; Constrained Longitudinal Data analysis with fixed effects for treatment, time, interaction of time by treatment, prior antihyperglycemic medication (monotherapy or dual therapy), and baseline eGFR (continuous)
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in the LSM vs. Glimepiride = -3.87, 95% CI 2-sided [-4.36 to -3.38]; [other analysis details as in outcome 5, analysis 1]

6. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) at Week 52 Excluding Rescue Approach
Description: This change from baseline reflects the Week 52 SBP minus the Week 0 SBP. Participants who met glycemic rescue criteria received open-label sitagliptin glycemic rescue medication.
Time Frame: Baseline and Week 52
Population: All randomized, treated participants with at least one SBP measurement (baseline or a post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
Number analyzed (Participants) | 448 | 440 | 437
mmHg | -2.25 [-3.36 to -1.13] | -3.81 [-4.91 to -2.71] | 0.95 [-0.15 to 2.06]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Glimepiride; Test type: Other; p < 0.001, Constrained Logitudinal Data Analysis; Difference in the LSM vs. Glimepiride = -4.77, 95% CI 2-sided [-6.29 to -3.25]; Constrained Logitudinal Data Analysis with fixed effects for treatment, time, interaction of time by treatment, prior anthyperglycemic medication (monotherapy or dual therapy), and baseline eGFR (continuous)
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Glimepiride; Test type: Other; p < 0.001, Constrained Logitudinal Data Analysis; Difference in the LSM vs. Glimepiride = -3.20, 0.001% CI 2-sided [-4.73 to -1.67]; [other analysis details as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Week 106
Description: The safety analysis population included all randomized participants who took at least one dose of trial treatment, 10 randomized participants from one trial site were excluded from these analyzes, and one randomized participant did not receive treatment.
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Glimepiride
All-Cause Mortality (participants affected / at risk) | 7/445 | 2/435 | 1/435
Serious Adverse Events (participants affected / at risk) | 41/445 | 32/435 | 30/435
Other Adverse Events (participants affected / at risk) | 110/445 | 104/435 | 165/435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=445) | Ertugliflozin 15 mg (N=435) | Glimepiride (N=435)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Atrial fibrillation aggravated (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Single vessel disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Triple vessel disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract aggravated (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Chorioretinal folds (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Senile cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ventral hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 1 (1)
Weakness generalised (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic calculous cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gangrene toe (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza A virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Purulent appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Recurrent urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sigmoid diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Knee ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Knee sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbosacral (joint) (ligament) sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Malleolar fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neck strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pertrochanteric fracture of femur, closed (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shoulder sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Calcifying tendinitis of shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in thigh (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Breast ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cancer of sigmoid colon (excl rectosigmoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metatypical basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid papillary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tubular adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Uterine fibroids (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Depression aggravated (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression worsened (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Recurrent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic retention of urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Choanal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Obstructive chronic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Foot ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic peripheral angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Leg ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=445) | Ertugliflozin 15 mg (N=435) | Glimepiride (N=435)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 12 (12) | 22 (24)
Common cold (Infections and infestations) | 21 (31) | 17 (29) | 23 (31)
Upper respiratory tract infection (Infections and infestations) | 27 (39) | 14 (19) | 18 (27)
Urinary tract infection (Infections and infestations) | 27 (30) | 28 (33) | 29 (36)
Asymptomatic hypoglycaemia (Metabolism and nutrition disorders) | 7 (11) | 4 (5) | 27 (87)
Hypoglycaemia (Metabolism and nutrition disorders) | 14 (31) | 25 (53) | 82 (470)
Headache (Nervous system disorders) | 25 (27) | 19 (22) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT01999218/Prot_SAP_000.pdf